CLINICAL TRIAL: NCT02269865
Title: Defining and Managing the Neuropsychological Abnormalities of Myotonic Dystrophy
Brief Title: Children's Health Research Institute(CHRI), Stanford Lucile Packard Children Hospital (LPCH) Protocol on Myotonic Dystrophy
Acronym: CHRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 28486
Record Dates: First submitted 2013-12-04; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Myotonic Dystrophy Type 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples and Cerebrospinal Fluid (CSF) samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Study to focus on the defining and managing the neuropsychological abnormalities of myotonic dystrophy and to find out if the neuropsychological abnormalities have any correlation with changes seen on Magnetic Resonance Imaging.

DETAILED DESCRIPTION:
Given the prevalence of DM, and assistance from The Myotonic Dystrophy Foundation (letter), we anticipate full recruitment of 8-17 year old subjects with DM1. The genetic counselor will help recruit 20 DM1 subjects, and 20 comparably aged controls, all of whom will complete MRI and neuropsychological tests. We anticipate full participation in evoked potential and blood tests, but estimate 30% will permit a lumbar puncture for CSF evaluation - done at the LPCH Ambulatory Procedure Unit with sedation as necessary. In total 40 MRIs will be done over 2 years, or 20 annually. Testing of Subjects

All neuropsychological evaluations will be performed in the morning in attempt to standardize wakefulness and stamina. Dr. Day's assessment of clinical status (~45 min) utilizes the Stanford myotonic dystrophy questionnaire, the University of Rochester MDHI, and the muscular impairment rating scale (MIRS)57, and records vital signs, current medications, spirometer, and disease history and progression. Given the frequency of sleep disorders in DM, subjects will complete the Affiliated Sleep Questionnaire, an online collection of extensive information in standardized format (see letter Dr. Mignot). After the clinical and neuropsychological assessments the subject and family members will have lunch prior to the MRI(75 min). In the mid-afternoon subjects will have evoked potentials in the Electrodiagnostics Lab(~90 min) followed by a lumbar puncture (if consenting) and blood draw in the LPCH APU(90 min). Subjects return home the same day, and Ms. Paulose contacts them several days later for feedback.

ELIGIBILITY:
Inclusion Criteria:

* 20 subjects with Myotonic Dystrophy type 1 aged 8 to 17 years and 20 controls who are healthy volunteers or siblings of affected subjects.

Exclusion Criteria:

-

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 20 subjects with Myotonic Dystrophy type 1 aged 8 to 17 years and 20 controls who are healthy volunteers or siblings of affected subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Define the neuropsychological abnormalities in Myotonic Dystrophy type 1 | 2 years
  The outcome of these studies will determine detailed spatial localization of white matter changes in DM1 children for the first time, and will establish a quantitative baseline with which future studies can determine the time course of the changes. The outcome results will determine whether functional abnormalities (fMRI, neuropsychological function, and evoked potentials) increase as white matter integrity deteriorates, and will explore tract-specific alteration of these effects. Defining cellular pathophysiology and CNS biomarkers of neurological dysfunction in DM will determine disease mechanisms and treatment pathways, and facilitate design of clinical and preclinical studies.

CONTACTS AND LOCATIONS:
Overall Officials: John W Day, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital, Stanford, Stanford, California, United States